CLINICAL TRIAL: NCT01987635
Title: Assessment of Sustained Systolic-to-diastolic Flexibility of the Mitral Valve Annulus With the Sorin MEMO 3D Mitral Anuloplasty Ring
Acronym: MEMO 3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/900
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Mitral Valve Disease
Keywords: Mitral valve disease; primarily regurgitation; necessitating surgical repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEMO 3D anuloplasty ring (Experimental): MEMO 3D anuloplasty ring
  Interventions: Device: MEMO 3D ring; Procedure: 3D Echocardiography
- rigid ring (Active Comparator): rigid ring
  Interventions: Device: Standard use of rigid ring.; Procedure: 3D Echocardiography

INTERVENTIONS:
Device: MEMO 3D ring — The experimental MEMO 3D ring is placed.
  Arms: MEMO 3D anuloplasty ring
Device: Standard use of rigid ring. — The rigid ring is placed, which is standard procedure.
  Arms: rigid ring
Procedure: 3D Echocardiography

SUMMARY:
Mitral valve reconstruction commonly requires the use of an anuloplasty device to assure long-term durability of the repair. Among mitral anuloplasty devices, varying from rigid to complete flexible ring substitutes, the most recent ones are aimed to restore the natural saddle shape of the mitral annulus, in order to decrease the stress tension on both mitral leaflets and chordal attachments. So far, even for flexible ring devices, the sustained flexibility of the device remained unproven, probably by cicatricial fibrotic tissue ingrowth after implantation.

Due to specific structural characteristics based on a nitinolstent with carbofilm-coating, the MEMO 3D ring device of SORIN claims preservation of the ring flexibility during the cardiac cyclus. Consequently, mitral anuloplasty with this device is expected to decrease the stress during the systolo-diastolic movements of the valve, and so, improve the late durability of the repair.

Echocardiography is the first-line technique for mitral valve assessment after surgical repair, for both intra-operative evaluation and serial follow-up of valve function. Recently, three-dimensional echocardiography has been introduced into clinical practice, affording qualitative and quantitative measurement of mitral valve function and size during the cardiac cycle.This method allows to quantify precisely the excursion of the mitral annulus between systole and diastole.

The aim of this study is to analyse the systolo-diastolic movement of the mitral annulus after the use of an anuloplasty with the SORIN MEMO 3D device, after surgical implantation and its sustainability, 1 year after implantation.

This hypothesis is tested in a case-controlled comparison with a standard used rigid ring device.

Therefore, 3-D echocardiography will be performed at the time of surgical repair, and after 1 year, to define the size and surface change of the mitral anuloplasty device during the cardiac cycle.

Based on a sample size calculation, 10 patients in each comparison group will be included, suggesting a study cohort of 20 patients eligible for mitral valve repair.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring the use of an mitral anuloplasty device to restore the mitral competence by surgery are potential candidates for study inclusion, if survival of at least more than 1 year is expected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01-16 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Difference of diameters and surface of the anuloplasty device between systolic and diastolic phase of the cardiac cycle in the MEMO 3D device, compared to another rigid ring device. | intra-operatively
  Difference of antero-posterior diameter, latero-lateral diameter and surface of the anuloplasty device between systolic and diastolic phase of the cardiac cycle in the MEMO 3D device, compared to another rigid ring device. The measurements are done with the use of 3-D echocardiography
Difference of diameters and surface of the anuloplasty device between systolic and diastolic phase of the cardiac cycle in the MEMO 3D device, compared to another rigid ring device. | 1 year after implantation.
  Difference of antero-posterior diameter, latero-lateral diameter and surface of the anuloplasty device between systolic and diastolic phase of the cardiac cycle in the MEMO 3D device, compared to another rigid ring device. The measurements are done with the use of 3-D echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Guy Vandenplas, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be